CLINICAL TRIAL: NCT02775747
Title: Platelet Rich Plasma Gel in Wound Closure in Recurrent Cesarean Section:Randomized Controlled Trial
Brief Title: PRP Gel in Wound Closure in Recurrent CS
Acronym: PRP-CS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, rasha medhat abdul-hady, Dr., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRP-CS
Record Dates: First submitted 2016-05-07; First posted 2016-05-18 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2016-04

CONDITIONS: Previous Incision; Scar; Previous Cesarean Section
MeSH Terms: conditions — Cicatrix | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- platelet rich plasma gel (Experimental): Injection of Platelet rich plasma (PRP) gel in 64 cases at time of wound closure in women undergoing cesarean section for improving wound healing after fullfit to all the inclusion and exclusion craiteria
  Interventions: Biological: platelet rich plasma gel
- Saline (Placebo Comparator): 64 Controlled Women with recurrent cesarean section and fullfit to all the inclusion and exclusion craiteria will reseve saline injection at time of wound closure
  Interventions: Biological: saline

INTERVENTIONS:
Biological: platelet rich plasma gel — Platelet rich plasma is prepared from fresh whole blood which is collected from a peripheral vein stored in acid citrare dextrose solution A (ACD-A)anticoagulant and processed to increase platelets by separating various components of blood
  Other Names: PRP; platelete rich plasma (PRP)
  Arms: platelet rich plasma gel
Biological: saline — 64 controlled women with recurrent cesarean section and fullfit to all inclusion and exclusion craiteria will reseve saline injection at time of wound closure
  Arms: Saline

SUMMARY:
There is limited application of the use of PRP in obstetrics, therefore there is a need for assessment if it is efficacy in improving skin wound healing in cesarean section.

DETAILED DESCRIPTION:
This study aims to assess the efficacy of injection of platelet rich plasma into the wound of recurrent cesarean section for improving wound healing and enhancing the shape of the wound in women undergoing cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* elective cesarean section
* Body mass index 18:25
* Hemoglobin more than 10.5 g/d
* Albumin within normal more than or equal 3.5 g/d

Exclusion Criteria:

* medical disorders(Diabetes mellitus,heart disease,hypertension,systemic lupus erythematosus)
* high risk pregnancy as (placenta previa,placenta accreta)
* patient on corticosteroids medication
* primigravida subjected cesarean section
* complicated cesarean section (increased operation time,blood transfusion, drain, scrubbing of multiple surgeons)
* cesarean section due to chorioaminionitis
* postoperative complication such as:postpartum hemorrhage, paralytic ileus, sever distention..) will be dropped out from the study

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Efficacy of PRP in Wound healing in cesarean section by 100 mm visual analog scale | one month
  Efficacy of PRP in Wound healing in cesarean section by 100 mm visual analog scale (VAS) for wound healing

SECONDARY OUTCOMES:
Assessment of the Cosmetic results of the wound by Modified Vancouver scar scale | one month
  Assessment of the Cosmetic results of the wound by Modified Vancouver scar scale

CONTACTS AND LOCATIONS:
Overall Officials: RASHA DR MEDHAT, MD, Principal Investigator — Ain Shams University; Rasha M Abdul-hady, MD, Principal Investigator — Ain Shams University
Locations (1):
- Rasha, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided